CLINICAL TRIAL: NCT05444712
Title: Transplantation After Complete Response In Patients With T-cell Lymphoma
Acronym: TRANSCRIPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL21_1095
Record Dates: First submitted 2022-06-08; First posted 2022-07-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: peripheral T-cell Lymphoma; autologous stem cell transplantation; chemotherapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): The chemotherapy is one of the following regimen administrated every 3 weeks for 6 cycles according to local investigator's choice based on usual practices and European Medical Agency (EMA) approval :
  * "Cyclophosphamide, doxorubicin, Vincristine and prednisone": (CHOP)
  * "Cyclophosphamide, doxorubicin, vincristine, etoposide and prednisone": (CHOEP)
  * "Brentuximab vedotin, cyclophosphamide, doxorubicin, prednisone": (BV-CHP) for ALCL lymphoma only (based on EMA approval)
  Interventions: Procedure: Chemotherapy + follow up
- Chemotherapy + ASCT (Active Comparator): Chemotherapy administrated every 3 weeks for 6 cycles according to local investigator's choice based on usual practices:
  Patients with ASCT strategy in Complete Response after 6 cycles will receive a High Dose Therapy (HDT) composed of BCNU, etoposide, cytarabine and melphalan (BEAM) as conditioning regimen before transplantation. That consolidation phase will lasts between 2 to 3 months
  Interventions: Procedure: Chemotherapy + ASCT + follow up

INTERVENTIONS:
Procedure: Chemotherapy + follow up — * Chemotherapy administrated every 3 weeks for 6 cycles according to local investigator's choice based on usual practices.
  * An intermediate evaluation will be performed after four cycles by PET-CT (or CT-Scan for non-avid PTCL)
  * A post-induction evaluation by PET-CT or CT-Scan will be done between 3 and 5 weeks after the last chemotherapy drug administration for all patients
  * A last evaluation by PET-CT or CT-Scan will be done between 08 and 12 weeks after the post-induction for all patients
  Arms: Chemotherapy
Procedure: Chemotherapy + ASCT + follow up — * Chemotherapy administrated every 3 weeks for 6 cycles according to local investigator's choice based on usual practices.
  * An intermediate evaluation will be performed after four cycles by PET-CT (or CT-Scan for non-avid PTCL)
  * The fifth or sixth cycles should be used as stem-cell mobilizing chemotherapy for patients with ASCT strategy
  * A post-induction evaluation by PET-CT or CT-Scan will be done between 3 and 5 weeks after the last chemotherapy drug administration for all patients
  * Patients with in Complete Response after 6 cycles will receive a High Dose Therapy as conditioning regimen before transplantation
  * A last evaluation by PET-CT or CT-Scan will be done between 08 and 12 weeks after the post-induction for all patients
  Arms: Chemotherapy + ASCT

SUMMARY:
Peripheral T-cell lymphoma (PTCL) encompasses a broad range of post-thymic (i.e., mature) sub-entities as defined by the 2017 WHO classification. The most common entities are angioimmunoblastic T-cell lymphoma (AITL) and other Tfh-phenotype PTCL or PTCL not otherwise specified (NOS), each representing approximately 20 to 25% of mature T- and NK/T-cell lymphomas. Compared to their B-cell counterparts, most PTCL confer dismal prognosis. In fact, except for anaplastic lymphoma kinase (ALK)-positive systemic anaplastic large cell lymphoma (sALCL), 10-year overall survival for patients with PTCL barely exceeds 30%. Given the infrequency and the heterogeneity of these malignancies, no real consensus on first-line treatment has been established for most PTCL.

The place of autologous stem cell transplantation (ASCT) as a consolidation procedure for patients with PTCL achieving a complete metabolic response after induction is still highly debated. ESMO recommendations and recent guidelines from a committee of the American Society for Blood and Marrow Transplantation currently propose ASCT as first-line therapy for transplant-eligible patients for all patients reaching at least a partial response (PR) after induction. NCCN guidelines (version 2.2017) recommend ASCT or observation in case of metabolic CR but salvage regimen in case of residual disease after induction.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years and < 70 years of age at the time of signing the informed consent form (ICF)
2. Patient fit enough to receive autologous stem cell transplant as a consolidation strategy as assessed by the local investigator
3. Hemoglobin level > 8g/dL (transfusion allowed); Neutrophil count >0.5 G/L; Platelets count > 50 G/L (transfusion allowed) Patient with histologically proven "nodal-type peripheral T-cell lymphoma (PTCL)" (latest WHO classification), not previously treated; as defined by the WHO classification, the following subtypes may be included,

   * PTCL, not otherwise specified
   * Follicular helper T-cell lymphomas: Angioimmunoblastic T-cell lymphoma and nodal PTCL with TFH phenotype and follicular T-cell lymphoma
   * Anaplastic large cell lymphoma, ALK-negative
4. Ann Arbor staging (I-IV) except stage I with normal LDH and PS<2 (i.e. stage I aaIPI 0)
5. Participant with a measurable disease by the Lugano criteria (i.e., longest diameter of a nodal site > 1.5 cm and/or longest diameter of an extranodal site > 1.0 cm and/or a hypermetabolic lesion)
6. FFPE Diagnostic tissue block should be available for central pathology review and ancillary molecular analyses
7. Participant with Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
8. Estimated minimum life expectancy of 3 months
9. Patient who understood and voluntarily signed and dated an informed consent prior to any study-specific assessments/procedures being conducted
10. Able to adhere to the study visit schedule and other protocol requirements
11. Patient covered by any social security system (France)
12. Patient who understands and speaks one of the country official languages
13. Males with partners of childbearing potential must agree to use effective birth control methods during the study as informed by the investigator in accordance with SmPC of each drugs administrated
14. Females of childbearing potential must agree to use effective birth control methods for at least 28 days before starting treatment; while participating in the study; during treatment interruptions and necessary period after the study as informed by the investigator in accordance with SmPC of each drugs administrated

Exclusion Criteria:

1. Known central nervous system or meningeal involvement by lymphoma
2. Impaired renal function (calculated MDRD or Cockcroft-Gault Creatinine Clearance < 30 ml/min) or impaired liver function tests (serum total bilirubin level > 2.0 mg/dl [34 µmol/L] (except in case of Gilbert's Syndrome, or documented liver or pancreatic involvement by lymphoma), serum transaminases (AST or ALT) > 3 upper normal limit unless they are related to the lymphoma.
3. The following types of T-cell lymphomas:

   * Adult T-cell lymphoma/leukemia (HTLV-1 related T-cell lymphoma)
   * Extranodal T-cell/NK-cell lymphoma, nasal type
   * Anaplastic large cell lymphoma, ALK-positive type
   * Cutaneous T cell lymphoma (mycosis fungoides, Sézary syndrome)
   * Primary cutaneous CD30+ T-cell lymphoproliferative disorder
   * Primary cutaneous anaplastic T-cell lymphoma
   * Enteropathy-associated T-cell lymphoma
   * Hepatosplenic T-cell lymphoma
   * Subcutaneous panniculitis-like T-cell lymphoma
   * Primary cutaneous gamma-delta T-cell lymphoma
   * Primary cutaneous CD8+ aggressive epidermotropic lymphoma
   * Primary cutaneous CD4+ small/medium T-cell lymphoma
4. Active malignancy other than the one treated in this research. Prior history of malignancies unless the patient has been free of the disease for ≥ 2 years. However, patients with the following history are allowed:

   1. Basal or squamous cell carcinoma of the skin
   2. Carcinoma in situ of the cervix
   3. Carcinoma in situ of the breast
   4. Incidental histologic finding of prostate cancer (T1a or T1b) using the tumor, nodes, metastasis clinical staging system
5. Vaccinated with live, attenuated vaccines within 6 months of enrollment
6. Use of any standard or experimental anti-cancer drug therapy before the start of treatment except COP (cyclophosphamide, vincristine, prednisone) in case of (or high risk of tumor lysis syndrome) or etoposide for a maximum of 3 doses (at a maximum dose of 150mg/m2) for HLH (Hemophagocytic Lymphohistiocytosis).
7. A corticosteroids therapy > 1mg/kg lasting more than 14 days prior to Cycle 1 Day 1
8. Positive serology for Human Immunodeficiency Virus (HIV) and Human T-Lymphotrophic Virus (HTLV1)

15. Active Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infections defined as:

* HBV :
* HBs Ag positive
* HBs Ag negative, anti-HBs antibody positive and anti-HBc antibody positive with detectable viral DNA
* HCV :

Anti-VHC antibody positive with detectable viral RNA 9. Pregnant, planning to become pregnant or lactating WOCBP 10. Any significant medical conditions, laboratory abnormality or psychiatric illness likely to interfere with the participation in this clinical study (according to the investigator's decision) 11. Person deprived of his/her liberty by a judicial or administrative decision 12. Person hospitalized without consent 13. Adult person under legal protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
to assess if ASCT is associated with a significant prolongation of progression-free survival (PFS) for patient with peripheral T-cell lymphoma (PTCL) reaching a complete response (CR) according to the response critter | When the last randomized patient has reached two years of follow-up or when 154 events (progression/relapse/new anti-lymphoma treatment/death) occured whichever comes first
  progression-free survival defined time from the date of randomization to the date of first documentation of relapse or progressive disease, death due to any cause, or receipt of subsequent systemic chemotherapy to treat residual or progressive peripheral T-cell lymphoma as determined by the investigator, whichever came first.

SECONDARY OUTCOMES:
Comparison of chemotherapy regimens + ASCT consolidation with chemotherapy regimens alone in terms of Overall survival (OS) | When the last randomized patient has reached two years of follow-up or when 154 events (progression/relapse/new anti-lymphoma treatment/death) occured whichever comes first
  Overall survival will be measured from the date of randomization to the date of death from any cause
Comparison of chemotherapy regimens + ASCT consolidation with chemotherapy regimens alone in terms of Overall response rate (ORR) and Complete Response Rate (CRR) | At the end of ASCT (8-12 weeks after post-induction evaluation)
  Overall Response Rate is defined as the proportion of subjects achieving best overall response of partial metabolic response (PMR) or complete metabolic response (CMR) at the end of ASCT (8-12 weeks after PIE). Assessment of response will be determined by investigator and based on Lugano Response Criteria 2014 (PET-CT-Based Response for FDG-avid lymphomas or CT-Based Response if not).
Comparison of chemotherapy regimens + ASCT consolidation with chemotherapy regimens alone in terms of duration of Response (DoR) | When the last randomized patient has reached two years of follow-up or when 154 events (progression/relapse/new anti-lymphoma treatment/death) occured whichever comes first
  Duration of response will be measured from the time of attainment of CMR or PMR to the date of first documented disease progression, relapse (based on investigator disease assessment), death from any cause or receipt of subsequent systemic chemotherapy to treat residual or progressive peripheral T-cell lymphoma as determined by the investigator, whichever came first.
Comparison of chemotherapy regimens + ASCT consolidation with chemotherapy regimens alone in terms of time to next Treatment (TTNT) | When the last randomized patient has reached two years of follow-up or when 154 events (progression/relapse/new anti-lymphoma treatment/death) occured whichever comes first
  TTNT will be measured from the date of randomization to the date of first documented administration of new anti-lymphoma treatment.
Comparison of chemotherapy regimens + ASCT consolidation with chemotherapy regimens alone in terms of quality of Life | When the last randomized patient has reached two years of follow-up or when 154 events (progression/relapse/new anti-lymphoma treatment/death) occured whichever comes first
  The EuroQol 5 Dimensions questionnaire (EQ5D-5L) will be administered at baseline and every three months during follow-up visit.
Comparison of chemotherapy regimens + ASCT consolidation with chemotherapy regimens alone in terms of cost-Effectiveness Analysis | When the last randomized patient has reached two years of follow-up or when 154 events (progression/relapse/new anti-lymphoma treatment/death) occured whichever comes first
  Will be expressed as the extra cost per a quality adjusted life year. To assess the mean cost per patient of each group, the number of resources consumed and the amounts refunded will be extracted from the French National Health Insurance Information System. The number of QALYs in each group of the trial will be assessed with survival time and the validated EuroQol 5 Dimensions questionnaire (EQ5D-5L).
Comparison of chemotherapy regimens + ASCT consolidation with chemotherapy regimens alone in terms of budget Impact Analysis | When the last randomized patient has reached two years of follow-up or when 154 events (progression/relapse/new anti-lymphoma treatment/death) occured whichever comes first
  budget impact analysis to assess the potential annual economic impact of the new management recommendation (with or without ASCL) for the French Public Health Insurance System across a 3-year time period.
Adjusted comparison of chemotherapy regimens (CHOP vs CHOEP) in non-sALCL in terms of Overall Response Rate (ORR) | at the end of induction (between 3 and 5 weeks after the last drug administration)
  Overall Response Rate is defined as the proportion of subjects achieving best overall response of partial metabolic response (PMR) at the end of induction. Assessment of response will be determined by investigator and based on Lugano Response Criteria 2014 (PET-CT-Based Response for FDG-avid lymphomas or CT-Based Response if not).
Adjusted comparison of chemotherapy regimens (CHOP vs CHOEP) in non-sALCL in terms of Complete Response rate (CRR) | at the end of induction (between 3 and 5 weeks after the last drug administration)
  complete metabolic response is defined as the proportion of subjects achieving complete metabolic response (CMR) at the end of induction. Assessment of response will be determined by investigator and based on Lugano Response Criteria 2014 (PET-CT-Based Response for FDG-avid lymphomas or CT-Based Response if not).
To evaluate the predictive value of total metabolic tumor volume (TMTV) on PET-CT | at patient enrollment
  Predictive value of TMTV on PET-CT
To Evaluate PET-CT Omics | at patient enrollment
  PET-Omics
The assessment of the early PET-CT predictive value after four cycles of chemotherapy on treatment response according to the IWC (International Workshop Criteria) Lugano 2014 | After four cycles of chemotherapy (each cycle is 3weeks)
  Predictive value of an early PET_CT after 4 cycles of chemotherapy on treatment response according to the IWC Lugano 2014

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel BACHY, Pr, Principal Investigator — HCL
Locations (48):
- France (48):
  - Chu D'Amiens - Hopital Sud, Amiens
  - Chu D'Angers, Angers
  - Ch Victor Dupouy, Argenteuil
  - Ch D'Avignon - Hopital Henri Duffaut, Avignon
  - Ch de La Cote Basque, Bayonne
  - Service d'Onco-radiolothérapie, Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Ch Metropole Savoie - Site Chambery, Chambéry
  - Chu Estaing, Clermont-Ferrand
  - Ch Alpes Leman, Contamine-sur-Arve
  - Hopital Henri Mondor, Créteil
  - René Olivier Casasnovas, Dijon
  - CHU Francois MITTERRAND, Dijon
  - Ch de Dunkerque, Dunkirk
  - Chd de Vendee, La Roche-sur-Yon
  - Ch de Versailles - Hopital Andre Mignot, Le Chesnay
  - CHU du Mans, Le Mans
  - Service Oncologie médicale, HOPITAL SAINT VINCENT-DE-PAUL, Lille
  - Service Hématologie Clinique et Thérapie Cellulaire, CHU DE LIMOGES - HOPITAL DUPUYTREN,, Limoges
  - Centre Leon Berard, Lyon
  - Chu de Montpellier, Montpellier
  - Chu de Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Chu de Nimes - Hopital Caremeau, Nîmes
  - Chr Orleans, Orléans
  - Hopital Cochin, Paris
  - Hopital de La Pitie Salpetriere, Paris
  - Hopital Necker, Paris
  - Hopital Saint Antoine, Paris
  - Ch de Perpignan, Perpignan
  - Chu de Bordeaux - Hopital Haut-Leveque, Pessac
  - Ch Perigueux, Périgueux
  - Chu Lyon-Sud, Pierre-Bénite
  - Ch Annecy Genevois, Pringy
  - Chu Pontchaillou_Rennes, Rennes
  - Ch de Roubaix - Hopital Victor Provo, Roubaix
  - Centre Henri Becquerel, Rouen
  - Service Hématologie, Institut Curie - Hôpital René HUGUENIN, Saint-Cloud
  - Chu de La Reunion - Hopital Felix Guyon, Saint-Denis
  - Chu de La Reunion - Ghsr, Saint-Pierre
  - Institut Cancerologie & Hematologie St-Etienne, Saint-Priest-en-Jarez
  - Ch de Saint-Quentin, Saint-Quentin
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer, Toulouse
  - Chu Bretonneau, Tours
  - Ch de Valence, Valence
  - Ch de Valenciennes - Hopital Jean Bernard, Valenciennes
  - Chu Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif